CLINICAL TRIAL: NCT00969228
Title: Immunogenicity, Reactogenicity and Safety Study to Evaluate Two Doses of the Lyophilised Formulation of the Human Rotavirus (HRV) Vaccine When Administered to Healthy Korean Infants Previously Uninfected With HRV
Brief Title: Study to Evaluate Immunogenicity, Reactogenicity and Safety of Rotarix™ Vaccine in Korean Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 112269; 2015-001545-81 (EudraCT Number)
Record Dates: First submitted 2009-08-20; First posted 2009-09-01 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Infections, Rotavirus; Rotavirus Vaccines
Keywords: Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rotarix Group (Experimental): Subjects received 2 oral doses of Rotarix according to a 0, 1 or 2-month schedule.
  Interventions: Biological: Rotarix ™
- Placebo Group (Placebo Comparator): Subjects received 2 oral doses of placebo according to a 0, 1 or 2-month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix ™ — Two oral doses
  Arms: Rotarix Group
Biological: Placebo — Two oral doses
  Arms: Placebo Group

SUMMARY:
The aim of this study is to assess the immunogenicity, reactogenicity and safety of the human rotavirus (HRV) Rotarix ™ vaccine when administered in healthy infants aged approximately 6-12 weeks at the time of first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 6 to 12 weeks of age at the time of the first dose of the vaccination.
* Written informed consent obtained from the parents or guardians of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a normal gestation period of between 37 and 41 weeks + 6 days inclusive.
* Subjects for whom the vaccination history is available from vaccination diary cards or medical charts.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine with the exception of the routine infant vaccines.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract or other serious medical condition as determined by the investigator.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Gastroenteritis (GE) within 7 days preceding the study vaccine administration.
* Previous confirmed occurrence of RV GE.
* Previous vaccination with rotavirus vaccine or planned use during the study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 684 (Actual)
Dates: Start 2009-08-25 (Actual); Primary Completion 2010-07-23 (Actual); Study Completion 2010-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- South Korea (11):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Goyang
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Iksan
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju Jeonbuk
  - GSK Investigational Site, Kwangju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=276

REFERENCES:
- [Background] Kim JS, Bae CW, Lee KY, Park MS, Choi YY, Kim KN, Kim JD, Park WS, Sin JB, Kim EA, Lee SG, Kim CS, Cha SH, Hong YJ, Shin SM, Shim GH, Choi KM, Yang JW, Liu A, Suryakiran PV, Han HH. Immunogenicity, reactogenicity and safety of a human rotavirus vaccine (RIX4414) in Korean infants: a randomized, double-blind, placebo-controlled, phase IV study. Hum Vaccin Immunother. 2012 Jun;8(6):806-12. doi: 10.4161/hv.19853. Epub 2012 Jun 1. PMID 22699440
- [Background] Kim JS et al. Assessment of immunogenicity, reactogenicity and safety of human rotavirus vaccine RIX4414 in Korean infants. Abstract presented at the Korean Society of Pediatric Infectious Diseases - 2011 Autumn Conference (KSPID). Seoul, S Korea, 12-15 November 2011.
- [Background] Buyse H, Vinals C, Karkada N, Han HH. The human rotavirus vaccine Rotarix in infants: an integrated analysis of safety and reactogenicity. Hum Vaccin Immunother. 2014;10(1):19-24. doi: 10.4161/hv.26476. Epub 2013 Oct 8. PMID 24047799
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 112269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112269 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotarix Group | Placebo Group
Started | 508 | 176
Completed | 465 | 162
Not Completed | 43 | 14
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Porcine circovirus detection in vaccine | 38 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 508 | 176 | 684
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.8 (1.25) | 8.9 (1.26) | 8.8 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231 | 79 | 310
  Male | 277 | 97 | 374

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for Anti-rotavirus Immunoglobulin A
Description: Seroconversion is defined as the appearance of antibodies with concentrations greater than or equal to 20 units per milliliter (U/mL) in the serum of subjects seronegative before vaccination.
Time Frame: One month after the second vaccine dose
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 318 | 114
subjects | 280 | 5

2. Secondary Outcome: Serum Anti-rotavirus Immunoglobulin A Antibody Concentrations
Description: Concentrations are given as Geometric Mean Concentrations (GMCs). Note: In the Placebo Group the value was below the assay cut-off (20 units per milliliter).
Time Frame: One month after the second vaccine dose
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: units per milliliter (U/mL)
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 280 | 114
units per milliliter (U/mL) | 208.5 [174.2 to 249.5] | NA [NA to NA] — Values were below the assay cut-off of 20 units per milliliter.

3. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited symptoms assessed include cough, diarrhoea, irritability, loss of appetite , fever and vomiting.
Time Frame: During the 8-day (Day 0 - Day 7) follow-up period after each vaccine dose.
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 508 | 176
subjects
  Cough | 180 | 66
  Diarrhoea | 20 | 7
  Irritability | 290 | 106
  Loss of appetite | 174 | 60
  Fever | 67 | 18
  Vomiting | 95 | 36

4. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Day 0 - Day 30) follow-up period after each vaccine dose
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 508 | 176
subjects | 148 | 59

5. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (2-3 months).
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 508 | 176
subjects | 17 | 13

6. Secondary Outcome: Number of Subjects Reporting Rotavirus Gastroenteritis Episode(s)
Time Frame: From Dose 1 up to 1 month after Dose 2.
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 508 | 176
subjects | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 8-day follow-up period after each dose of vaccine. Unsolicited adverse events: during the 31-day follow-up after any dose of Rotarix vaccine or placebo. Serious adverse events: during the entire study period (2-3 months)
Arm/Group | Rotarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 17/508 | 13/176
Other Adverse Events (participants affected / at risk) | 367/508 | 134/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=508) | Placebo Group (N=176)
Bronchiolitis (Infections and infestations) | 6 | 5
Gastroenteritis (Infections and infestations) | 5 | 4
Pyrexia (General disorders) | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia apiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Solitary kidney (Congenital, familial and genetic disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=508) | Placebo Group (N=176)
Cough (General disorders) | 180 | 66
Irritability (General disorders) | 290 | 106
Loss of appetite (General disorders) | 174 | 60
Fever (General disorders) | 67 | 18
Vomiting (General disorders) | 95 | 36
Nasopharynigitis (Infections and infestations) | 29 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.